CLINICAL TRIAL: NCT05316584
Title: A Novel Remote Patient and Medication Monitoring Solution to Improve Adherence and PerSiStence With Inflammatory Bowel DiSease Therapy-ASSIST Study
Brief Title: A Novel Remote Patient and Medication Monitoring Solution to Improve Adherence and PerSiStence With IBD Therapy
Acronym: ASSIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Vanderbilt University Medical Center (Other); New York University (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sandra Quezada, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22010339
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory bowel disease; Crohn disease; Ulcerative colitis; Adherence; Remote monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to blind participants to their respective group assignment. However, to minimize bias, we will collect all outcome data electronically by study staff at the Data Management Center at the University of North Carolina masked to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring (Experimental): At the time of a medication dose, participants scan the smart label by tapping it with their mobile device. Participants receive a notification on their device indicating that their medication adherence was updated. Each day a medication is due, patients receive a morning reminder through SMS message notifying them on their medications schedule. If patients fail to scan the label at a given time (as expected by their specific medication regimen), they will receive an end of day text message. Participants will also complete a patient reported outcome (PRO) 2 assessment at baseline, and then monthly for the entire 12 months of the study through an HTML link sent to patients by SMS message. If nonadherence is present and/or moderate to severe symptoms, an alert will be triggered to the research team. The research team can send the PRO2 survey to patients at any given time, at their discretion, if patients are experiencing a flare or at the time of a change in medication dose.
  Interventions: Behavioral: Remote monitoring
- Control (No Intervention): The standard of care for participants in this study is modeled after the standard of care at all five study sites. Standard of care is based on current evidence-based guidelines including a comprehensive assessment, a guideline-concordant therapy plan, scheduled and as needed clinic visits, scheduled and as needed telephone calls, and administration of educational fact sheets about disease-specific topics when appropriate. Personnel used to provide standard of care at each site will vary and may include nurse coordinators, advanced practice providers, social workers, psychologists, dieticians, pharmacists, and other ancillary staff.

INTERVENTIONS:
Behavioral: Remote monitoring — See prior description of the intervention.
  Arms: Remote Monitoring

SUMMARY:
The investigators hypothesize that use of a remote monitoring digital health system that supports medication taking and monitoring of symptoms will improve adherence, clinical outcomes, and decrease healthcare utilization compared to standard care in participants with inflammatory bowel disease initiating oral or subcutaneous treatment. The investigators are conducting a 12-month, multicenter, randomized, controlled trial to assess the feasibility and effectiveness of a remote monitoring digital health system on adherence, clinical outcomes, and healthcare utilization.

The investigators will address the following specific aims:

1. Compare adherence as measured by the medication possession ratio in participants using a remote monitoring digital health system compared to standard of care.
2. Compare clinical outcomes and healthcare utilization in participants using a remote monitoring digital health system compared to standard of care.

DETAILED DESCRIPTION:
The investigators hypothesize that use of a remote monitoring digital health system that supports medication taking and monitoring of symptoms will improve adherence, clinical outcomes, and decrease healthcare utilization compared to standard care in participants with inflammatory bowel disease (IBD) initiating oral or subcutaneous treatment. The investigators are conducting a 12-month multicenter, randomized, controlled trial to assess the feasibility and effectiveness of a remote monitoring digital health system on adherence, clinical outcomes, and healthcare utilization.

Adult participants with IBD with regular access to a mobile device or tablet initiating therapy with an oral or subcutaneous treatment for IBD at one of the five sites will be eligible to participate. Participants will be randomized 2:1 to the intervention or standard care. Eligible participants will complete an informed consent and baseline survey gathering demographic and clinical information.

TapptTM digital health system (developed by Synchronyx) is a remote therapeutic monitoring and digital engagement solution that monitors real-time medication adherence patterns through smart label technologies, capture patient reported outcomes (PROs) and barriers to care, and process patient data through algorithms that trigger personalized digital and human touchpoints between clinical visits. The research team will input information into the system on the intervention participant's medication to be tracked, dose, and frequency of dosing. Participants in the intervention group will be shipped the smart labels to be affixed to the pill bottle, pen, or syringe of the newly prescribed medication. Prior to receiving their medication, participants will receive virtual training on how to attach and use the proprietary labels, set up their participant profile, use the participant-facing web app, and seek technical helpdesk support. At the time of a medication dose, participants will scan the label by tapping it with their mobile device to verify that they are taking the medication. Upon scanning, participants immediately will receive a notification on their device indicating that the label was successfully scanned, and that their medication adherence was updated in their profile. The app offers participants visibility into their medication adherence patterns and upcoming doses, as well as the opportunity to respond to in-app questions that capture barriers towards adherence, IBD symptoms, and patient report outcomes (PROs). This information will also be available to the research and clinical team in real-time via the provider dashboard. Most importantly, the dashboard's artificial intelligence-based algorithm will send email alerts to the clinical team if participant's adherence, symptoms, or PROs fall below predetermined thresholds. For oral medications, mean adherence <86% in a 2-week period will trigger an alert. For SC medications, an alert will be generated if a dose is 10 days late for administration. A PRO 2 score for UC or CD of 2 or more will trigger an alert. If alerts are triggered for non-adherence, a clinical nurse, pharmacist, or social worker will contact the participant to identify barriers to adherence; remediation will be initiated if possible.

The primary outcome of the proposed study will be the difference in mean medication possession ratio (MPR) between the intervention and control group during the 12-month study. Secondary outcomes will include self-reported adherence (MARS-5), clinical response and remission (Harvey Bradshaw Index for CD and partial Mayo score of UC), steroid-free response and remission, PROMIS measures of Fatigue, Sleep Disturbance, Pain Interference, Anxiety, Depression, and Quality of Life, self-efficacy (IBD Self-Efficacy Scale), new steroid use, and health care utilization (urgent care or emergency room visit, unplanned office visit, hospitalization, and/or surgery).

Assuming 2 intervention participants for every 1 control with an adherence rate among controls of 0.65 and 0.9 in intervention participations with a Type 1 error rate of 0.05 and power of 0.9, we will need to enroll 82 intervention participants and 41 controls (n=123). All analyses will be completed using intention to treat principles. For categorical variables, the groups will be compared using the Chi Square test (Fisher's Exact if not normally distributed). For continuous variables, the groups will be compared using t tests (Wilcoxon signed rank if not normally distributed). We will also build logistic and linear regression models to adjust for confounding variable for the outcomes of interest. Possible confounding variables include but are not limited to route of administration, gender, insurance type, disease type, age, concurrent psychiatric disease, smoking, and concurrent steroid and/or narcotic use.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Have documented IBD based on usual diagnostic criteria including clinical symptoms and findings from endoscopy, radiology studies, and histology
3. Initiating treatment with a new oral or subcutaneous treatment for IBD
4. Have access to a mobile smartphone (iPhone 7 or later; Android release date 2012 or later) with reliable data and/or Wi-Fi access
5. Ability to understand the protocol and provide informed consent in English

Exclusion Criteria:

1. Inability to speak and read English
2. Inability to comply with the study protocol
3. Presence of an ileostomy, colostomy, ileoanal pouch anastomosis, or ileorectal anastomosis
4. Patients initiating oral corticosteroids only (without concurrent use of an oral or subcutaneous maintenance therapy)
5. Imminent surgery (within the next 60 days)
6. History of short bowel syndrome
7. Uncontrolled medical or psychiatric disease at the opinion of the investigator

   1. Degenerative neurologic condition
   2. Unstable angina
   3. Symptomatic peripheral vascular disease
   4. Malignancy within the last 2 years (excluding squamous or basal cell cancers of the skin)
   5. Poorly controlled depression, mania, and schizophrenia
   6. Serious active infection requiring antimicrobial therapy (excluding CD patients with perianal CD on antibiotics)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 1 year
  Medication possession ratio
Self-reported medication adherence | 1 year
  MARS-5, scores from 5 to 25 with higher scores indicated greater adherence

SECONDARY OUTCOMES:
Healthcare utilization | 1 year
  Rates of healthcare utilization including office and ER visits, hospitalizations, and diagnostic testing
IBD Disease activity | 1 year
  Harvey Bradshaw Index ( for participants with Crohn's disease only), minimum score 0, no maximum score, higher scores indicated greater disease activity
IBD Disease activity (objective) | 1 year
  C reactive protein, minimum value 0, no maximum value, higher values indicate greater disease activity
Patient Reported Outcomes, Quality of Life | 1 year
  PROMIS Global Health, T scores from 0-100, 50 is the population mean, higher scores indicate better quality of life
Self-efficacy | 1 year
  IBD Self-efficacy scale, scores range from 29-290 with higher scores indicated greater self-efficacy
IBD Disease Activity | 1 year
  Simple clinical colitis activity index (participants with ulcerative colitis only), minimum score 0, maximum score 19, higher scores indicate greater disease activity
IBD Disease Activity (objective) | 1 year
  Fecal calprotectin, minimum value 0, no maximum value, higher values indicate greater disease activity
IBD Disease Activity (objective) | 1 year
  Mayo Endoscopic score (participants with ulcerative colitis only), minimum score 0, maximum score 3, higher scores indicate greater disease activity
IBD Disease Activity (objective) | 1 year
  Simple endoscopic score (participants with Crohn's disease only), minimum score 0, maximum score 60, higher scores indicate greater disease activity
Patient Reported Outcome (Pain interference) | 1 year
  PROMIS Pain Interference, T scores from 0-100, 50 is the population mean, higher scores indicate more pain
Patient Reported Outcome (Anxiety) | 1 Year
  PROMIS Anxiety, T scores from 0-100, 50 is the population mean, higher scores indicate more anxiety
Patient Reported Outcome (Depression) | 1 year
  PROMIS Depression, T scores from 0-100, 50 is the population mean, higher scores indicate more depression
Patient Reported Outcome (Fatigue) | 1 year
  PROMIS Fatigue, T scores from 0-100, 50 is the population mean, higher scores indicate more fatigue
Patient Reported Outcome (Sleep Disturbance) | 1 year
  PROMIS Sleep Disturbance, T scores from 0-100, 50 is the population mean, higher scores indicate more sleep disturbance

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - New York University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
After publication, raw data will be made available to other investigators upon receipt of a written request. Release of datasets to secondary users will be subject to approval by the investigators. The request must include a reason for review of the data and type of dataset they wish to receive, and a copy of a curriculum vitae. The dataset provided will be deidentified to prevent breach of confidentiality. Investigators requesting to review our data must sign an agreement that they will not attempt to obtain protected health information on participants. In addition to the raw data, investigators will receive a list of variable and coding definitions. The agreement will specify, the data are to be used for IRB-approved research purposes only and data will not be transferred to other users by the recipient. The methodology for the Tappt system and for the proposed trial will be published.
Time Frame: See above
Access Criteria: See above

REFERENCES:
- [Derived] Axelrad J, Long M, Horst S, Afzali A, Sapir T, Fajardo K, De Felice K, Sandler R, Cross R. A Novel Remote Patient and Medication Monitoring Solution to Improve Adherence and Persistence With Inflammatory Bowel Disease Therapy (ASSIST Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Dec 15;11(12):e40382. doi: 10.2196/40382. PMID 36520519